CLINICAL TRIAL: NCT03472976
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of Inactivated Influenza A/H5N1 Vaccine Administered Intradermally With or Without Topical Aldara(R) in Healthy Young Adults
Brief Title: H5N1 With or Without Topical Aldara in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-0050; HHSN272201300015I
Record Dates: First submitted 2018-03-15; First posted 2018-03-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2018-08-14

CONDITIONS: Avian Influenza; Influenza Immunisation
Keywords: Healthy Young Adults; Immunogenicity; Inactivated Influenza A/H5N1 Vaccine; Phase I Clinical Trial; Reactogenicity; Safety; Topical Aldara(R)
MeSH Terms: conditions — Influenza in Birds; Influenza, Human | interventions — Imiquimod; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): 0.1 ml of influenza A/H5N1 IIV vaccine (9 mcg HA) intradermally 15 minutes after the application of approximately 250 mg of Imiquimod (Aldara) cream topically (deltoid) on Day 1 and Day 22. N=25
  Interventions: Drug: Imiquimod; Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Vietnam/1203/04
- Group 2 (Experimental): 0.1 ml of influenza A/H5N1 IIV vaccine (9 mcg HA) intradermally 15 minutes after the application of approximately 250 mg of Aqueous Cream B.P. (Control Cream) topically (deltoid) on Day 1 and Day 22. N=25
  Interventions: Other: Aqueous Cream B.P.; Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Vietnam/1203/04

INTERVENTIONS:
Other: Aqueous Cream B.P. — Aqueous Cream B.P. will be used as the control cream. An equivalent of 250mg of the cream will be applied and rubbed into the skin until it vanishes, on the deltoid area 5-15 minutes prior to vaccine administration.
  Arms: Group 2
Drug: Imiquimod — Aldara (imiquimod 5%) cream is an immune response modifier for topical administration. 250 mg of the cream, equivalent to 12.5 mg of imiquimod will be applied and rubbed into the skin until it vanishes, on the deltoid area 5-15 minutes prior to vaccine administration.
  Arms: Group 1
Biological: Influenza Virus Vaccine, Monovalent A/H5N1 A/Vietnam/1203/04 — Inactivated monovalent subvirion H5N1 vaccine containing hemagglutinin (HA) of A/Vietnam/1203/04

SUMMARY:
Phase I randomized, double-blind, placebo-controlled trial in 50 males and non-pregnant females, 18 to 49 years old, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of inactivated A/H5N1 influenza vaccine administered intradermally (ID) with topical Aldara or control cream as a 2-dose regimen. The vaccine will be administered using the MicronJet600(TM) device. Subjects will be assigned to 2 treatment arms (25 subjects per treatment arm). Group A will receive two doses of A/H5N1 IIV ID with pre-application of topical Aldara on Days 1 and 22. Group B will receive two doses of A/H5N1 IIV ID with pre-application of topical control cream on Days 1 and 22. The duration of this study will be approximately 20 months with patient participation duration approximately 7 months. The primary objectives of this study are: 1) to assess the safety and reactogenicity after 2 doses of A/H5N1 IIV vaccine containing 9 mcg HA per dose administered ID approximately 21 days apart with topical Aldara or control cream; 2) to assess the serum HAI antibody responses 21 days after receipt of the 2nd dose of A/H5N1 IIV administered ID at 9 mcg HA per dose with topical Aldara or control cream.

DETAILED DESCRIPTION:
This is a Phase I randomized, double-blind, placebo-controlled trial in 50 males and non-pregnant females, 18 to 49 years old, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of inactivated A/H5N1 influenza vaccine administered intradermally (ID) with topical Aldara or control cream as a 2-dose regimen. The vaccine will be administered using the MicronJet600(TM) device. Subjects will be assigned randomly to 1 of 2 treatment arms (25 subjects per treatment arm) to receive 2 doses of A/H5N1 IIV administered ID with topical Aldara or control cream. Group A will receive two doses of A/H5N1 IIV (9 mcg HA/dose) ID with pre-application of topical Aldara on Days 1 and 22. Group B will receive two doses of A/H5N1 IIV (9 mcg HA/dose) ID with pre-application of topical control cream on Days 1 and 22. The duration of this study will be approximately 20 months with patient participation duration approximately 7 months. The primary objectives of this study are: 1) to assess the safety and reactogenicity after 2 doses of A/H5N1 IIV vaccine containing 9 mcg HA per dose administered ID approximately 21 days apart with topical Aldara or control cream; 2) to assess the serum HAI antibody responses 21 days after receipt of the 2nd dose of A/H5N1 IIV administered ID at 9 mcg HA per dose with topical Aldara or control cream. The secondary objectives are: 1) to assess unsolicited non-serious adverse events (AEs) following receipt of 2 doses of A/H5N1 IIV administered ID approximately 21 days apart with topical Aldara or control cream; 2) to assess medically-attended adverse events (MAAEs) including new-onset chronic medical conditions (NOCMCs), and potentially immune mediated medical conditions (PIMMCs) following receipt of two doses of A/H5N1 IIV administered ID approximately 21 days apart with topical Aldara or control cream for six months after last vaccination; 3) to assess the serum neutralizing (Neut) antibody responses 21 days following receipt of the 1st and 2nd dose of A/H5N1 IIV administered ID with topical Aldara or control cream; 4) to assess the serum HAI antibody responses 21 days following receipt of the 1st dose of A/H5N1 IIV administered ID with topical Aldara or control cream; 5) to assess the serum HAI and Neut antibody responses 7 days following receipt of the 2nd dose of A/H5N1 IIV administered ID with topical Aldara or control cream.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, 18 to 49 years old, inclusive.
4. Are in good health, as determined by vital signs (oral temperature, pulse, and blood pressure), medical history, and physical examination to ensure any existing medical diagnoses or conditions (except those exclusionary) are stable.

   - Stable chronic medical condition - no change in prescription medication, dose, or frequency of medication in the last 2 months (defined as 60 days) and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months (defined as 180 days). Any change that is due to change of health care provider, insurance company etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a violation of this inclusion criterion.

   -- Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity. Note: Topical, nasal, and inhaled medications (with the exception of steroids as outlined in the Subject Exclusion Criteria), vitamins, and contraceptives are permitted.
5. Oral temperature is less than 100.0 degrees F.
6. Pulse is 47 to 100 bpm, inclusive.
7. Systolic blood pressure is 85 to 150 mm Hg, inclusive.
8. Diastolic blood pressure is 55 to 95 mmHg, inclusive.
9. Women of childbearing potential must use an acceptable method of contraception from 30 days prior to vaccination until 60 days after the last study vaccination.

   - Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year of the last menses if menopausal).

   -- Includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with a vasectomized partner, male condoms with the use of applied spermicide, intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill"). Method of contraception will be captured on the appropriate data collection form.
10. Female subjects of childbearing potential must have a negative urine pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination.

   - An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation.

   - Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.
3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
4. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma skin cancers that are not active are permitted.
5. Have known HIV, chronic hepatitis B virus, or chronic hepatitis C infection.
6. Have known hypersensitivity or allergy to eggs, egg or chicken protein, or other components of the study vaccine.
7. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
8. Have a history of Guillain-Barré Syndrome.
9. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
10. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
11. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
12. Have taken oral or parenteral (including intraarticular) corticosteroids of any dose within 30 days prior to study vaccination.
13. Have taken high-dose dose inhaled corticosteroids within 30 days prior to study vaccination.

    - High-dose defined as the dose in mcg/day of an inhaled steroid used alone or in combination with other inhaled medications. Available at: https://www.nhlbi.nih.gov/health-pro/guidelines/current/asthma-guidelines/quick-reference-html#estimated-comparative-daily-doses

    -- Topical and nasal steroids are permissible.
14. Received any licensed live vaccine within 30 days prior to the first study vaccination.
15. Received a licensed inactivated vaccine within 14 days prior to the first study vaccination.
16. Plans to receive any licensed vaccine from the time of the first study vaccination through the follow-up visit at approximately 21 days after the last study vaccination.
17. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
18. Received an experimental agent within 30 days prior to the first study vaccination, or expects to receive an experimental agent during study paticipation.

    - Including vaccine, drug, biologic, device, blood product, or medication.

    -- Other than from participation in this study.
19. Are participating or plan to participate in another clinical trial with an interventional agent that will be received during study participation.

    -Including agent (licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) during the 7-month study period.
20. Prior participation in a clinical trial of influenza A/H5 vaccine or have a history of A/H5 actual or potential exposure or infection prior to the first study vaccination.

    - Assigned to a group receiving influenza A/H5 vaccine (does not apply to documented placebo recipients)
21. Plan to travel outside the U.S. (continental U.S., Hawaii and Alaska) in the time between the first study vaccination and 21 days after the last study vaccination.
22. Female subjects who are breastfeeding.
23. Blood donation or planned blood donation within 30 days prior to the study vaccination through 30 days after the last blood drawn for this study.
24. Have signs or symptoms that could confound or confuse assessment of study vaccine reactogenicity.

    - The study vaccination should be postponed/deferred until signs or symptoms have resolved and if within the acceptable protocol-specified window for that visit.
25. Receiving or planning to receive Aldara, imiquimod or resiquimod for any clinical indication during the duration of study participation.
26. Patients with autoimmune skin diseases such as psoriasis or atopic dermatitis.
27. Known allergy to Aldara or its components, and/or to aqueous cream B.P.

    - Methyl hydroxybenzoate (E 218) and propyl hydroxybenzoate (E 216) may cause allergic reactions (possibly delayed). Cetyl alcohol and stearyl alcohol may cause local skin reactions (e.g. contact dermatitis).

    -- Liquid paraffin, white soft paraffin, cetostearyl alcohol, sodium lauryl sulfate, phenoxyethanol may cause local skin reactions (e.g. contact dermatitis).
28. Presence of large or dark tattoos on the deltoid area that would significantly interfere with reactogenicity assessment.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) of serum HAI antibodies | Day 1
Geometric mean titers (GMTs) of serum HAI antibodies | Day 43
Occurrence of all SAEs | Day 1 through Day 202
Occurrence of solicited injection site AEs | Day 1 through Day 8
Occurrence of solicited injection site AEs | Day 22 through Day 29
Occurrence of solicited systemic AEs | Day 1 through Day 8
Occurrence of solicited systemic AEs | Day 22 through Day29
Occurrence of study vaccine-related SAEs | Day 1 through Day 202
Percentage of subjects achieving a serum HAI antibody titer of 40 or greater against the A/H5N1 antigen contained in the study vaccine | Day 43
Percentage of subjects achieving HAI seroconversion against study vaccine (pre-vaccination HAI titer <10 and post-vaccination HAI titer > / = 40 or pre-vaccination HAI titer > / =10 and a min 4-fold rise in post-vaccination HAI antibody titer | Day 43

SECONDARY OUTCOMES:
GMT of serum HAI antibody against the A/H5N1 antigen contained in the study vaccine | Day 22
GMT of serum Neut antibody against the A/H5N1 antigen contained in the study vaccine | Day 1
GMT of serum Neut antibody against the A/H5N1 antigen contained in the study vaccine | Day 22
GMT of serum Neut antibody against the A/H5N1 antigen contained in the study vaccine | Day 43
Occurrence of all unsolicited non-SAEs | Day 1 through Day 43
Occurrence of Medically-Attended Adverse Events (MAAEs), including New-Onset Chronic Medical Conditions (NOCMCs) and Potentially Immune-Mediated Medical Conditions (PIMMCs) | Day 1 through Day 202
Occurrence of study vaccine-related unsolicited non-serious AEs | Day 1 through Day 43
Percentage of subjects achieving a serum HAI antibody titer of 40 or greater against the A/H5N1 antigen contained in the study vaccine | Day 22
Percentage of subjects achieving a serum Neut antibody titer of 40 or greater against the A/H5N1 antigen contained in the study vaccine | Day 1
Percentage of subjects achieving a serum Neut antibody titer of 40 or greater against the A/H5N1 antigen contained in the study vaccine | Day 22
Percentage of subjects achieving a serum Neut antibody titer of 40 or greater against the A/H5N1 antigen contained in the study vaccine | Day 43
Percentage of subjects achieving HAI seroconversion against the A/H5N1 antigen contained in the study vaccine | Day 22
Percentage of subjects achieving Neut seroconversion (pre-vaccination Neut titer < 10 and post-vaccination Neut titer > / = 40 or pre-vaccination Neut titer > / = 10 and a min 4-fold rise in post-vaccination Neut antibody titer) | Day 22
Percentage of subjects achieving Neut seroconversion (pre-vaccination Neut titer < 10 and post-vaccination Neut titer > / = 40 or pre-vaccination Neut titer > / = 10 and a min 4-fold rise in post-vaccination Neut antibody titer) | Day 43
Proportion of subjects with GMT of serum Neut antibody against the A/H5N1 antigen contained in the study vaccine | Day 29
Proportion of subjects with seroconversion against the A/H5N1 antigen contained in the study vaccine | Day 29
Proportion of subjects with titer of 40 or greater of serum HAI antibody against the A/H5N1 antigen contained in the study vaccine | Day 29
Proportion of subjects with titer of 40 or greater of serum Neut antibody against the A/H5N1 antigen contained in the study vaccine | Day 29
Secondary Proportion of subjects with GMT of serum HAI antibody against the A/H5N1 antigen contained in the study vaccine | Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas, United States

REFERENCES:
- [Derived] El Sahly HM, Atmar RL, Sendra E, Wegel A, Keitel WA. Topical Imiquimod Does Not Provide an Adjuvant Effect When Administered With Inactivated Influenza A/H5N1 Vaccine in Healthy Young Adults. J Infect Dis. 2021 Nov 22;224(10):1712-1719. doi: 10.1093/infdis/jiab206. PMID 33852718